CLINICAL TRIAL: NCT05163925
Title: A Prospective Single Center Study to Evaluate Safety and Efficacy of the EUROSETS Extracorporeal Membrane Oxygenation ECMOLIFE SYSTEM in Clinical Extracorporeal Life Support Applications EUROSETS ECMO STUDY
Brief Title: EUROSETS ECMO Study in Clinical Extracorporeal Life Support Applications
Status: Recruiting | Type: Observational
Sponsor: Eurosets S.r.l. (Industry)
Responsible Party: Sponsor
Other Study IDs: ECMO Study CIP 4.0_07.03.2025
Record Dates: First submitted 2021-09-24; First posted 2021-12-20 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-03

CONDITIONS: Extracorporeal Membrane Oxygenation Complication
Keywords: Extracorporeal Life Support Applications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Laboratory values pre-ECLS and daily during ECLS support
  * Hemoglobin
  * Hematocrit
  * Leukocytes
  * Platelets
  * Creatinine
  * BUN (Blood Urea Nitrogen)
  * AST (Aspartate-Aminotransferase)
  * ALT (Alanine-Aminotransferase)
  * Gamma GT (Gain of Thyroid)
  * LDH (Lactate Dehydrogenase)
  * Bilirubin
  * C-reactive protein
  * Hemolysis index
  * Fibrinogen
  * D-dimer if applicable
  * aPTT (activated partial Thromboplastin Time) or anti-Xa if applicable
  * Activated clotting time if applicable
  * Lactate
  * pH (acid base indicator)
  * pO2 (Oxygen partial pressure)
  * pCO2 (Carbon dioxide partial pressure)
  * SO2 (Oxygen saturation)
  * HCO3 (Bicarbonate)
  * BE (Base Excess)
  * SvO2 (Mixed venous oxygen saturation) if applicable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EUROSETS ECMOLIFE SYSTEM: Thirty consecutive patients that require ECLS and who receive the EUROSETS ECMOLIFE SYSTEM will be included. ECMOLIFE System is a perfusion system enabling operation and monitoring of extracorporeal circulation. ECMOLIFE System operates, powers, controls and regulates ECMOLIFE Centrifugal Pump which represents the disposable blood pump. ECMOLIFE System, when used in combination with ECMOLIFE Centrifugal Pump, is suitable for full or partial cardiac, circulatory and pulmonary support.
  ECMOLIFE System is composed by an active programmable console (ECMOLIFE Console), a bearing-less motor driver (ECMOLIFE Motor driver), and sensors for blood parameters detection (flow rate, pressure, temperature, SvO2 and Hb). The console is equipped with an integrated back-up which in case of primary unit failure may be operated in combination with a back-up motor driver and flowmeter (besides, the ECMOLIFE system includes an Heater cooler device).
  Interventions: Device: Eurosets ECMO Life System

INTERVENTIONS:
Device: Eurosets ECMO Life System — ECMOLIFE System in combination with ECMOLIFE Centrifugal Pump and ECC (extra-corporeal-circulation) Tubing Set is intended to pump blood through the extracorporeal circuit to provide extracorporeal circulation.
  ECMOLIFE System must be used only in combination with ECMOLIFE Centrifugal Pump.
  ECMOLIFE System is intended to operate in the following hospital environments: Operating Room, Catheter Laboratory, Emergency Room, Intensive Care Unit and during intra-hospital patient transportation from one to another Unit.
  ECMOLIFE System is intended to be used by qualified healthcare professionals specifically trained in the field of extracorporeal circulation: Perfusionists (Thoracic Cardiovascular Surgery - OR), Intensivists, ICU Nurses (ICU), Emergency physicians / Intensivists (ER), Cardiologist (CathLab).

SUMMARY:
This is a prospective single-center study designed for evaluation of safety and performance of the Conformitè Europëenne (CE)-marked EUROSETS ECMOLIFE SYSTEM, composed by: ECMOLIFE console, ECMO TUBING SET, ECMO OXYGENATOR and ECMOLIFE CENTRIFUGAL PUMP, HEATER COOLER (called ECMOLIFE HC) in all clinical ECLS applications (e.g. post-cardiotomy ECLS as well as application for cardiogenic shock after myocardial infarction or resulting from other etiologies, as well as ECLS application in patients under cardiopulmonary resuscitation (eCPR) and protected PCI) in 30 consecutive patients.

All demographic and perioperative variables (ECMOLIFE SYSTEM -related and unrelated ECLS complications, performances of the ECMOLIFE SYSTEM) will be analyzed. Surgical techniques will be recorded. Follow-up information on survival and any adverse cardiac and cerebrovascular events will be gathered routinely by outpatient clinic and telephone calls until 30 days after ECLS initiation or hospital discharge.

DETAILED DESCRIPTION:
The prevalence of post-cardiotomy extracorporeal life support (PC-ECLS) varies between 0.6% and 3.6% of all cardiac surgical cases and represents one of the most common applications of ECLS. While a majority of patients can be weaned from cardiopulmonary bypass using inotropic and vasoactive medication, some experience refractory cardiac and/or pulmonary dysfunction requiring prolonged postoperative mechanical circulatory support. Veno-arterial extracorporeal membrane oxygenation (VA-ECMO) support is a respected therapeutic option for short-term mechanical circulatory support in these critically ill patients. Indications for PC-ECLS usually include intra-operative failure to wean from cardiopulmonary bypass due to perioperative left, right or biventricular failure, or refractory cardiogenic shock/cardiac arrest in the postoperative period. While ECLS can be a life-saving therapy, it is characterized by a high mortality and morbidity due to neurologic and vascular complications amongst others.

Recently published studies reported that long-term prognosis of in-hospital survivors after ECMO support following cardiovascular surgery remains unsatisfactory, however, patients who survive have the chance to make a full recovery despite a very unfavorable prognosis without VA-ECMO. Predisposing risk factors influencing long-term survival are not fully known, however this knowledge is necessary for adequate patient selection and comprehensive decision-making prior to ECMO implantation in order to identify those patients who will truly benefit from ECMO support, since unrestrained use might disproportionately increase hospital costs and consume valuable resources.

Recently, the Extracorporeal Life Support Organization (ELSO) Registry reported a remarkable increase in the use of ECLS as a supportive therapy after cardiac surgery. However, a disappointing trend was observed with regards to the in-hospital survival rate, reaching only 15% in the latest period.

Despite this increase in use and new technological developments in this area, only a few comprehensive and dedicated reports about PC-ECLS have been presented. Nevertheless, PC-ECLS has represented the main indication for ECLS utilization and is characterized by specific aspects (duration and type of underlying disease, severity of comorbidities, indication and type of surgical procedure, modality of access and timing of implant, complication types and rates) when compared to other ECLS indication Cardiovascular diseases (CVD) are responsible for more than 4 million deaths in Europe per year. Thereby, CVD account for approximately 45% of mortality in Europe. Apart from medical and ethical aspects, this poses an economical disaster: annual costs of roughly 210 trillion USD. Among cardiovascular diseases, coronary heart disease alone is responsible for 1 million deaths per year. Myocardial infarction (MI) is often the initial manifestation of coronary heart disease, caused by myocardial ischemia and necrosis leading to an acute decrease of cardiac function. Clinically, patients in cardiogenic shock present hypotensive, unresponsive to intravenous fluid challenge and with clinical and laboratory signs of critical end organ malperfusion requiring pharmacologic and/or mechanical circulatory support.

Cardiogenic shock (CS) is the leading cause of death after myocardial infarction and occurs in 5-10% of all cases of MI. Trials such as SHOCK, IABP-SHOCK II and IMPRESS in Severe Shock all revealed a one-year mortality of approximately 50%, which reflects constant mortality rates over the last 20 years, in spite of the applied therapeutic strategies and devices.

The unacceptably high mortality and morbidity in CS is an unsolved clinical problem despite all available treatment options.

Protected PCI is the application of Mechanical Circulatory Support (MCS) during percutaneous coronary intervention in high-risk patients, meaning that in such cases MCS systems are implanted prophylactically despite hemodynamic stability to avoid deleterious complications. The overall patient condition and temporary impairment based on the acute situation of an underlying myocardial infarction or coronary ischemia, without a manifested cardiogenic shock, are potential reasons for a "prophylactic" use of MCS.

Due to the increasing complexity of procedures and patients, feasibility of such interventions is becoming more dependent on the availability of MCS, in order to guarantee hemodynamic support during revascularization. Safety and outcome of such high-risk PCIs can potentially be improved by the application of MCS and the onset of complications such as arrhythmias, hemodynamic instability and related complications during the procedure can be reduced.

In Patient without ROSC (return of spontaneous circulation) during CPR, reestablishment of circulation by emergent VA-ECLS implantation may be indicated, since eCPR is able to improve the outcome of patients after prolonged resuscitation and no-ROSC scenario.

In 2019, at the Medical University of Vienna 25 patients were treated with eCPR (approximately 9% of all CPR-patients), 20 of these patients after OHCA (out of hospital cardiac arrest). Five patients (20%) survived with a good neurologic outcome.

In the eCPR setting, time between circulatory arrest and its recovery by the ECMO circuit, is a major crucial and impacting factor as well. The ease of use in terms of device implantation would be of high importance in those cases in particular.

In summary, for every indication, devices used in ECLS require maximum reliability and must be able to generate adequate flow for full circulatory support and minimize blood trauma especially in the setting of prolonged support. Additionally, handling and monitoring should be non-complicated, the need for frequent patient transports (operating room - ICU - remote hospital facilities as required) should be taken into account. New devices should be evaluated considering these factors- next to assessment of outcome and device-related and unrelated ECLS complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years
* VA-ECLS application using the EUROSETS ECMOLIFE SYSTEM (e.g. cardiogenic shock, post cardiotomy low cardiac output syndrome, cardiac arrest, high risk percutaneous coronary intervention, eCPR)

Exclusion Criteria:

* Patients <18 years
* Pregnant and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty consecutive patients that require ECLS and who receive the EUROSETS ECMOLIFE SYSTEM will be included. As the current study is a prospective study, choice of the device is based on surgeons' preference. ECLS usually is an unplanned procedure, post-hoc informed consent will be obtained in ECLS survivors before hospital discharge. However, when a patient clearly stated in the patient file he or she does not wish to participate in any trials, this will be honored. A screening log providing detailed information on inclusion or reasons for exclusion will be kept in record.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Rate of Device Malfunction | in-hospital, 30 days
  Rate of device malfunction of the EUROSETS device (ECMOLIFE console, ECMO TUBING SET, ECMO OXYGENATOR and ECMOLIFE CENTRIFUGAL PUMP, HEATER COOLER (called ECMOLIFE HC)) of total patients enrolled.
Rate of device related complications | in-hospital, 30 days
  Rate of device related complications of the EUROSETS device (ECMOLIFE console, ECMO TUBING SET, ECMO OXYGENATOR and ECMOLIFE CENTRIFUGAL PUMP, HEATER COOLER (called ECMOLIFE HC)) of total patients enrolled.

SECONDARY OUTCOMES:
Rate of Mortality | in-hospital, 30 days
  Rate of in-hospital and 30 day mortality.
Rate of Adverse Events | in-hospital, 30 days
  Rate of in-hospital and 30 day adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Petralia, Dott., Study Director — Eurosets S.r.l.
Locations (1):
- Medical University of Vienna, Department of Cardiac Surgery, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rastan AJ, Dege A, Mohr M, Doll N, Falk V, Walther T, Mohr FW. Early and late outcomes of 517 consecutive adult patients treated with extracorporeal membrane oxygenation for refractory postcardiotomy cardiogenic shock. J Thorac Cardiovasc Surg. 2010 Feb;139(2):302-11, 311.e1. doi: 10.1016/j.jtcvs.2009.10.043. PMID 20106393
- [Background] Elsharkawy HA, Li L, Esa WA, Sessler DI, Bashour CA. Outcome in patients who require venoarterial extracorporeal membrane oxygenation support after cardiac surgery. J Cardiothorac Vasc Anesth. 2010 Dec;24(6):946-51. doi: 10.1053/j.jvca.2010.03.020. PMID 20599396
- [Background] Whitman GJ. Extracorporeal membrane oxygenation for the treatment of postcardiotomy shock. J Thorac Cardiovasc Surg. 2017 Jan;153(1):95-101. doi: 10.1016/j.jtcvs.2016.08.024. Epub 2016 Aug 31. PMID 27666787
- [Background] Smedira NG, Blackstone EH. Postcardiotomy mechanical support: risk factors and outcomes. Ann Thorac Surg. 2001 Mar;71(3 Suppl):S60-6; discussion S82-5. doi: 10.1016/s0003-4975(00)02626-6. PMID 11265868
- [Background] Saxena P, Neal J, Joyce LD, Greason KL, Schaff HV, Guru P, Shi WY, Burkhart H, Li Z, Oliver WC, Pike RB, Haile DT, Schears GJ. Extracorporeal Membrane Oxygenation Support in Postcardiotomy Elderly Patients: The Mayo Clinic Experience. Ann Thorac Surg. 2015 Jun;99(6):2053-60. doi: 10.1016/j.athoracsur.2014.11.075. Epub 2015 Apr 10. PMID 25865760
- [Background] Fukuhara S, Takeda K, Garan AR, Kurlansky P, Hastie J, Naka Y, Takayama H. Contemporary mechanical circulatory support therapy for postcardiotomy shock. Gen Thorac Cardiovasc Surg. 2016 Apr;64(4):183-91. doi: 10.1007/s11748-016-0625-4. Epub 2016 Feb 13. PMID 26874519
- [Background] Sauer CM, Yuh DD, Bonde P. Extracorporeal membrane oxygenation use has increased by 433% in adults in the United States from 2006 to 2011. ASAIO J. 2015 Jan-Feb;61(1):31-6. doi: 10.1097/MAT.0000000000000160. PMID 25303799
- [Background] McCarthy FH, McDermott KM, Kini V, Gutsche JT, Wald JW, Xie D, Szeto WY, Bermudez CA, Atluri P, Acker MA, Desai ND. Trends in U.S. Extracorporeal Membrane Oxygenation Use and Outcomes: 2002-2012. Semin Thorac Cardiovasc Surg. 2015 Summer;27(2):81-8. doi: 10.1053/j.semtcvs.2015.07.005. Epub 2015 Jul 22. PMID 26686427
- [Background] Townsend N, Wilson L, Bhatnagar P, Wickramasinghe K, Rayner M, Nichols M. Cardiovascular disease in Europe: epidemiological update 2016. Eur Heart J. 2016 Nov 7;37(42):3232-3245. doi: 10.1093/eurheartj/ehw334. Epub 2016 Aug 14. No abstract available. PMID 27523477
- [Background] Timmis A, Townsend N, Gale C, Grobbee R, Maniadakis N, Flather M, Wilkins E, Wright L, Vos R, Bax J, Blum M, Pinto F, Vardas P; ESC Scientific Document Group. European Society of Cardiology: Cardiovascular Disease Statistics 2017. Eur Heart J. 2018 Feb 14;39(7):508-579. doi: 10.1093/eurheartj/ehx628. PMID 29190377
- [Background] Timmis A, Townsend N, Gale CP, Torbica A, Lettino M, Petersen SE, Mossialos EA, Maggioni AP, Kazakiewicz D, May HT, De Smedt D, Flather M, Zuhlke L, Beltrame JF, Huculeci R, Tavazzi L, Hindricks G, Bax J, Casadei B, Achenbach S, Wright L, Vardas P; European Society of Cardiology. European Society of Cardiology: Cardiovascular Disease Statistics 2019. Eur Heart J. 2020 Jan 1;41(1):12-85. doi: 10.1093/eurheartj/ehz859. PMID 31820000
- [Background] Harjola VP, Lassus J, Sionis A, Kober L, Tarvasmaki T, Spinar J, Parissis J, Banaszewski M, Silva-Cardoso J, Carubelli V, Di Somma S, Tolppanen H, Zeymer U, Thiele H, Nieminen MS, Mebazaa A; CardShock Study Investigators; GREAT network. Clinical picture and risk prediction of short-term mortality in cardiogenic shock. Eur J Heart Fail. 2015 May;17(5):501-9. doi: 10.1002/ejhf.260. Epub 2015 Mar 28. PMID 25820680
- [Background] van Diepen S, Katz JN, Albert NM, Henry TD, Jacobs AK, Kapur NK, Kilic A, Menon V, Ohman EM, Sweitzer NK, Thiele H, Washam JB, Cohen MG; American Heart Association Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Quality of Care and Outcomes Research; and Mission: Lifeline. Contemporary Management of Cardiogenic Shock: A Scientific Statement From the American Heart Association. Circulation. 2017 Oct 17;136(16):e232-e268. doi: 10.1161/CIR.0000000000000525. Epub 2017 Sep 18. PMID 28923988
- [Background] Hochman JS, Sleeper LA, Webb JG, Sanborn TA, White HD, Talley JD, Buller CE, Jacobs AK, Slater JN, Col J, McKinlay SM, LeJemtel TH. Early revascularization in acute myocardial infarction complicated by cardiogenic shock. SHOCK Investigators. Should We Emergently Revascularize Occluded Coronaries for Cardiogenic Shock. N Engl J Med. 1999 Aug 26;341(9):625-34. doi: 10.1056/NEJM199908263410901. PMID 10460813
- [Background] Thiele H, Zeymer U, Neumann FJ, Ferenc M, Olbrich HG, Hausleiter J, Richardt G, Hennersdorf M, Empen K, Fuernau G, Desch S, Eitel I, Hambrecht R, Fuhrmann J, Bohm M, Ebelt H, Schneider S, Schuler G, Werdan K; IABP-SHOCK II Trial Investigators. Intraaortic balloon support for myocardial infarction with cardiogenic shock. N Engl J Med. 2012 Oct 4;367(14):1287-96. doi: 10.1056/NEJMoa1208410. Epub 2012 Aug 26. PMID 22920912
- [Background] Thiele H, Schuler G, Neumann FJ, Hausleiter J, Olbrich HG, Schwarz B, Hennersdorf M, Empen K, Fuernau G, Desch S, de Waha S, Eitel I, Hambrecht R, Bohm M, Kurowski V, Lauer B, Minden HH, Figulla HR, Braun-Dullaeus RC, Strasser RH, Rochor K, Maier SK, Mollmann H, Schneider S, Ebelt H, Werdan K, Zeymer U; IABP-SHOCK II Trial Investigators. Intraaortic balloon counterpulsation in acute myocardial infarction complicated by cardiogenic shock: Design and rationale of the Intraaortic Balloon Pump in Cardiogenic Shock II (IABP-SHOCK II) trial. Am Heart J. 2015 Apr;169(4):e7-8. doi: 10.1016/j.ahj.2015.01.009. Epub 2015 Jan 30. No abstract available. PMID 25819870
- [Background] Ouweneel DM, Eriksen E, Sjauw KD, van Dongen IM, Hirsch A, Packer EJ, Vis MM, Wykrzykowska JJ, Koch KT, Baan J, de Winter RJ, Piek JJ, Lagrand WK, de Mol BA, Tijssen JG, Henriques JP. Percutaneous Mechanical Circulatory Support Versus Intra-Aortic Balloon Pump in Cardiogenic Shock After Acute Myocardial Infarction. J Am Coll Cardiol. 2017 Jan 24;69(3):278-287. doi: 10.1016/j.jacc.2016.10.022. Epub 2016 Oct 31. PMID 27810347
- [Background] Schober A, Sterz F, Herkner H, Wallmueller C, Weiser C, Hubner P, Testori C. Emergency extracorporeal life support and ongoing resuscitation: a retrospective comparison for refractory out-of-hospital cardiac arrest. Emerg Med J. 2017 May;34(5):277-281. doi: 10.1136/emermed-2015-205232. Epub 2017 Feb 17. PMID 28213587
- [Background] Poppe M, Schriefl C, Steinacher A, Clodi C, Warenits AM, Nurnberger A, Hubner P, Holzer M, Horvat J, Wiedemann D, Weiser C. Extracorporeal cardiopulmonary resuscitation at the emergency department: A retrospective patient selection evaluation. Eur J Anaesthesiol. 2020 Apr;37(4):280-285. doi: 10.1097/EJA.0000000000001142. PMID 31860604
- [Background] Ouweneel DM, Schotborgh JV, Limpens J, Sjauw KD, Engstrom AE, Lagrand WK, Cherpanath TGV, Driessen AHG, de Mol BAJM, Henriques JPS. Extracorporeal life support during cardiac arrest and cardiogenic shock: a systematic review and meta-analysis. Intensive Care Med. 2016 Dec;42(12):1922-1934. doi: 10.1007/s00134-016-4536-8. Epub 2016 Sep 19. PMID 27647331
- [Background] Wengenmayer T, Rombach S, Ramshorn F, Biever P, Bode C, Duerschmied D, Staudacher DL. Influence of low-flow time on survival after extracorporeal cardiopulmonary resuscitation (eCPR). Crit Care. 2017 Jun 22;21(1):157. doi: 10.1186/s13054-017-1744-8. PMID 28637497